CLINICAL TRIAL: NCT02842788
Title: Prospective Study on the Prevalence on the Use of Prone Positioning in ARDS Patients
Brief Title: Prevalence of Prone Positioning Use in ARDS Patients
Acronym: APRONET
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0468
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: prone position; acute respiratory distress syndrome (ARDS); mechanical ventilation; ICU; prevalence
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARDS patients receiving invasive mechanical ventilation in ICU: 1. ARDS criteria (Berlin definition) fulfilled the day of the study, whatever the ARDS stage. The onset of ARDS could have been established at any time between ICU admission and study day but ARDS criteria must be still present the day of the study. The ARDS criteria are listed below
     * Within 1 week of a known clinical insult or new or worsening respiratory symptoms
     * Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules
     * Respiratory failure not fully explained by cardiac failure or fluid overload. Need objective assessment (eg, echocardiography) to exclude hydrostatic edema if no risk factor present
  2. PaO2/FIO2 ≤ 300 with Positive end-expiratory pressure (PEEP) ≥ 5 cmH2O
  3. Age ≥ 18 years
  4. Intubated or tracheotomized and mechanically ventilated
  Interventions: Procedure: Prone positioning

INTERVENTIONS:
Procedure: Prone positioning — Turning the patient face down for several consecutive hours

SUMMARY:
Prone positioning has been shown to improve survival in patients with acute respiratory distress syndrome (ARDS). However, a recent large observational study found that prone positioning was used in only 7% of all ARDS patients, and 16% in the severe category. However, this study did not focus on the prone position per se. In present study, the investigators would like to explore the rate of use of prone positioning in ARDS patients and the reasons why this treatment was not applied. The present study is one-day prevalence study repeated four times over one year.

The hypothesis is that the rate of use of prone position is greater than 50% in the severe ARDS category.

ELIGIBILITY:
Inclusion Criteria:

* 1.ARDS criteria (Berlin definition) fulfilled the day of the study, whatever the ARDS stage. The onset of ARDS could have been established at any time between ICU admission and study day but ARDS criteria must be still present the day of the study. The ARDS criteria are listed below

  * Within 1 week of a known clinical insult or new or worsening respiratory symptoms
  * Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules
  * Respiratory failure not fully explained by cardiac failure or fluid overload. Need objective assessment (eg, echocardiography) to exclude hydrostatic edema if no risk factor present
* 2.PaO2/FIO2 ≤ 300 with PEEP ≥ 5 cmH2O
* 3.Age ≥ 18 years
* 4.Intubated or tracheotomized and mechanically ventilated

Exclusion Criteria:

* Patient non intubated the day of the study
* No criteria for ARDS the day of the study even if these criteria were present between ICU admission and day of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS under mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 736 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of the use of the prone position in ARDS | Day 1
  Number of patients with ARDS receiving prone position divided by number of patients with ARDS on the day of the study

SECONDARY OUTCOMES:
Prevalence of the use of the prone position in each ARDS category | Day 1
  Number of patients with ARDS in each category receiving prone position divided by number of patients with ARDS in each category on the day of the study
Occurence of reasons for not using prone position in ARDS patients | Day 1
  Reasons: No severe hypoxemia for the clinician, Intracranial hypertension, Mean arterial pressure < 65 mmHg, Unstable fractures, Pneumothorax with previous single drain, External cardiac stimulation or internal pacemaker inserted for less than 48 hours, Tracheotomy for less than 15 days (not for access to airways for the current mechanical ventilation purpose), Severe facial trauma or facial surgery in the last 15 days, Sternotomy in the last 15 days, Venous thrombosis treated by anticoagulant molecule for less than 48 hours, Massive hemoptysis requiring interventional radiology or other emergency procedure, Pregnant woman, Excess in workload, Other reason
PaO2 | Day 1
  oxygenation (PaO2) to assess the physiological response to the prone position session
PaO2/FIO2 | Day 1
  oxygenation (PaO2/FIO2) to assess the physiological response to the prone position session
Duration of prone position session | Day 1
  Difference between time of onset to time of end (consecutive hours)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Guérin, Pr, Principal Investigator — Réanimation médicale, Hôpital de la Croix Rousse, CHU de Lyon, France
Locations (1):
- Réanimation médicale, Hôpital de la Croix Rousse, CHU de Lyon, France, Lyon, France